CLINICAL TRIAL: NCT00385931
Title: A Multi-centre Study to Evaluate the Effects of Valsartan and the Combination of Valsartan and Simvastatin on Blood Pressure (Ambulatory and Std Cuff) and on Biochemical Markers of Endothelial Function (hsCRP, MCP-1, Serum F2 Isoprostanes, PAI-1, tPA, PICP, PIIINP, MMP9, MMP1, TIMP 1), Safety and Tolerability
Brief Title: Efficacy and Safety of Valsartan and the Combination of Valsartan and Simvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAS489A2301
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Hypertension; Hypercholesterolemia; Dyslipidemia
Keywords: Hypertension; high cholesterol; valsartan; simvastatin
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Dyslipidemias | interventions — Valsartan; Simvastatin

INTERVENTIONS:
Drug: Valsartan and simvastatin

SUMMARY:
This study will assess and compare the efficacy and safety of valsartan and the combination of valsartan and simvastatin in patients with high blood pressure and high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 50 years of age
* Mild to moderate essential systolic hypertension (grades 1 and 2 WHO classification) defined as MSSBP ≥ 150 mmHg and <180mmHg
* Simultaneous primary hypercholesterolemia or mixed dislipidemia (Fredrickson Types IIa and IIb) defined by LDL-C level ≥ 130 mg/dL and <190 mg/dL and triglyceride levels ≤ 400 mg/dL despite dietary therapy
* Off medication at randomization

Exclusion Criteria:

* Severe hypertension (grade 3 WHO classification
* ≥ 180 mm Hg systolic or ≥ 110 mm Hg (diastolic)
* secondary form of hypertension
* known Keith-Wagener Grade III or IV hypertensive retinopathy
* history of hypertensive encephalopathy or cerebrovascular accident within the preceding 12 months
* transient ischemic cerebral attack during the preceding 6 months
* dyslipidemia secondary to other causes
* Type 1 diabetes mellitus
* Type 2 diabetes mellitus with poor glucose control
* history of systemic inflammatory diseases
* serum CK more than twice ULN
* sodium depletion
* malignancy in preceding 5 years history of heart failure
* myocardial infarction within the preceding 12 months
* second or third degree heart block
* concomitant refractory angina pectoris
* symptomatic arrhythmia
* valvular heart disease
* Any condition/surgery that may alter absorption, distribution, metabolism, excretion of any drug (e.g. history of major gastrointestinal tract surgery, inflammatory bowel syndrome, pancreatic dysfunction, impaired renal or liver function)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2002-01; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ambulatory systolic blood pressure at 12 weeks

SECONDARY OUTCOMES:
Change from baseline at 12 weeks for ambulatory diastolic blood pressure, systolic and diastolic blood pressure (std cuff), day and nighttime blood pressures, biochemical markers of endothelial function & lipid levels
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States